CLINICAL TRIAL: NCT03091699
Title: The Acute Effects of Moderate Intensity Exercise and Nicotine on Cognition in Smokers
Brief Title: Effects of Exercise and Nicotine on Cognition in Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Professor/Director of the Exercise Health and Psychology Lab, Western University, Canada
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Exercise and Nicotine
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Smoking Cessation
Keywords: Smoking; Nicotine; Exercise; Cognition
MeSH Terms: conditions — Smoking Cessation; Smoking; Motor Activity | interventions — Nicotine; Tobacco Products

STUDY DESIGN:
Intervention Model Description: Sequential two stage trial. Stage 1 will utilize a within-counterbalanced approach while stage 2 will utilize a randomized trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate intensity exercise (Experimental): The Exercise intervention will persist of a 20-minute bout of moderate intensity aerobic exercise which by definition is 40-65% of Maximum Heart Rate. Exercise consisted of a 2-minute warm-up, followed by 15 min of walking at a rate, which will allow you to reach 2/3 of your max heart rate, and then a 3-minute cool down on a treadmill equaling 20 minutes. Heart Rate will be examined with Polar Wearlink coded Heart Rate monitors to attain the specific exercise intensity.
  Interventions: Behavioral: Moderate Intensity Exercise
- Nicotine Inhalation (Active Comparator): The nicotine inhalation group will smoke a cigarette to completion of their choice, in the 20 minute time period allocated in the Exercise and Health Psychology Lab psychological assessment room (the room will be equipped with windows that allow for ventilation and an air purifier. During this time the participant will refrain from conversation.
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Participants will be required to smoke a cigarette to completion in a 20 minute time frame.
  Other Names: Cigarettes
  Arms: Nicotine Inhalation
Behavioral: Moderate Intensity Exercise — Participants will be required to perform 20 minutes of acute moderate intensity exercise (brisk walk) on a treadmill.
  Arms: Moderate intensity exercise

SUMMARY:
Adult smokers will participate in a two stage testing trial, where the first stage will utilize a within-subject counterbalance design and individuals will participate in both conditions. The second stage will utilize a two-arm randomized control trail. The two conditions are (a) moderate intensity exercise and (b) nicotine inhalation. The primary measure of assessment will be reaction time and accuracy on the N-back task.

DETAILED DESCRIPTION:
The burden of smoking tobacco on the Canadian public is well-documented. Typically, two thirds of Canadian smokers will consider a quit attempt over the next six months. When an individual who is addicted to nicotine stops administering the psycho-stimulate cognitive deficits and tobacco cravings arise and are at the forefront of an unsuccessful quit attempt. Studies have shown that smoking or nicotine administration enhances alerting and orienting attention, short-term episodic memory, and working memory in smokers who were deprived or minimally deprived of nicotine. Moderate intensity exercise has been shown to increase many cognitive functions of the brain in non-smokers. Moderate intensity exercise also has been shown to increase cognition more than nicotine in a non-smoking population. Research regarding the effects of moderate exercise on cognition of non- deprived, as well as nicotine- deprived smokers is unknown.

The study will begin in April of 2017. The main purpose of this project is to examine if exercise could be a pragmatic alternative to smoking in cognitive deficits that arise during a quit attempt.

Thirsty four adult smokers will follow the protocol listed below:

Stage I will utilize a within subjects counter-balanced design. Previous to arrival for phase I participants will be asked to keep consumption of coffee to half a cup the day of testing, abstain from alcohol and drugs for at least 18 hours prior to testing, and smoke a cigarette of choice 30 minutes prior to arrival (for standardization). Participants will be urged to arrive at the same time for each visit. Upon arrival to the Exercise and Health Psychology lab (located in room 408 of the Arthur and Sonia Labatt Health Science Building at Western University) participants will be verified as smokers (based on the reading from the piCO+ Smokerlyzer being greater than 10 P.P.M.), given the letter of information and sign the informed consent form. Participants will also be asked to complete a demographic survey, smoking history questionnaire, PAR-Q readiness for exercise, Godin Leisure-Time Exercise Questionnaire, Fagerstrom Test for Nicotine Dependence, and pre nicotine or pre exercise questionnaire. Vitals (heart rate and blood pressure) will be assessed following the completion of the questionnaires as well as post intervention in the seated position. Prior to evaluation on the N-back task (cognitive memory task described below) a practice stage with be conducted until the participant can consistently score 75% or higher on three consecutive trials to eliminate a learning effect. After establishing familiarity a baseline cognition score will be conducted. The subject will then be given a 5 minute break (i.e., to use the lavatory). Following the break the participants will be randomized into either the exercise or nicotine inhalation group. The interventions are as followed; Moderate Intensity Exercise will persist of a 20-minute bout of moderate intensity aerobic exercise. Exercise consisted of a 2-minute warm-up, followed by 15 min of walking at a rate, which will allow you to reach 2/3 of your max heart rate, and then a 3-minute cool down on a treadmill equaling 20 minutes. The Nicotine inhalation group will smoke a cigarette to completion of their choice, in the 20 minute time period allocated. During this time the participant will refrain from conversation. The post intervention assessment will begin within two minutes of the completion of either intervention. The second visit of phase I will take place the following day at the same time (if possible). During the second visit the participant's will complete the pre nicotine or pre exercise questionnaire and vitals will be monitored pre and post intervention. The participants will participate in the intervention that they have not received on the first visit (for example, if the participant received nicotine inhalation on the first visit the participant will receive moderate intensity aerobic exercise on the second visit). Within two minutes of completion the post treatment N-back task assessment will begin. Previous to arrival for stage II participants will be asked to keep consumption of coffee to half a cup the day of testing, abstain from alcohol and drugs for at least 18 hours prior to testing, and to abstain from smoking for at least 12 hours (overnight abstinence). Stage II will utilize the same participants as phase I but they will be examined in a nicotine-deprived state (12 hours) for baseline N-back scores and then randomized into nicotine inhalation group or exercise treatment group where post intervention N-back scores will be obtained. Pre nicotine or pre exercise questionnaire will be completed and vitals (heart rate and blood pressure) will be assessed pre and post intervention. Smoking abstinence will be validated with the piCO+ Smokerlyzer reading being less than 10 P.P.M.

This study will (a) provide information about the cognition of non-deprived smokers and nicotine deprived smokers (b) demonstrate if moderate intensity exercise would be a pragmatic alternative to nicotine for replenishing working memory deficits in these populations (c) add to the literature on moderate intensity exercise being a valid aid for smokers attempting a real quit attempt (d) assist in the development of new cessation programs involving exercise.

ELIGIBILITY:
Inclusion Criteria:

* Fit the criteria of a smoker (smoke more than 5 cigarettes a day and on baseline assessment blow greater than 10 P.P.M. analyzed with the piCO+ Smokerlyzer.
* At least 18 years old
* Physically able to perform exercise
* Read and write in English
* Must have an email or telephone for communication

Exclusion Criteria:

* COPD or inhaler dependent
* Recent health issues such as a heart attack
* Participants taking prescription medication for depression or asthma
* Pregnant
* Unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Cognition (working memory) accuracy | 1 day
  intervention effects on the 3-back task accuracy (percentage of correct responses)
Cognition (working memory) reaction time | 1 day
  intervention effects on the 3-back task reaction time (milliseconds)

SECONDARY OUTCOMES:
Cognition (working memory) accuracy | 1 day
  intervention effects on the 0,1,2-back task and accuracy (percentage of correct responses)
Cognition (working memory) reaction time | 1 day
  intervention effects on the 0,1,2-back task and accuracy (percentage of correct responses)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, PhD, Principal Investigator — Professor
Locations (1):
- Western University, London, Ontario, Canada

REFERENCES:
- [Background] Heishman SJ, Kleykamp BA, Singleton EG. Meta-analysis of the acute effects of nicotine and smoking on human performance. Psychopharmacology (Berl). 2010 Jul;210(4):453-69. doi: 10.1007/s00213-010-1848-1. Epub 2010 Apr 24. PMID 20414766
- [Background] Hughes JR. Effects of abstinence from tobacco: etiology, animal models, epidemiology, and significance: a subjective review. Nicotine Tob Res. 2007 Mar;9(3):329-39. doi: 10.1080/14622200701188927. PMID 17365765
- [Background] Jonides J, Schumacher EH, Smith EE, Lauber EJ, Awh E, Minoshima S, Koeppe RA. Verbal Working Memory Load Affects Regional Brain Activation as Measured by PET. J Cogn Neurosci. 1997 Jul;9(4):462-75. doi: 10.1162/jocn.1997.9.4.462. PMID 23968211
- [Background] Stolz D, Scherr A, Seiffert B, Kuster M, Meyer A, Fagerstrom KO, Tamm M. Predictors of success for smoking cessation at the workplace: a longitudinal study. Respiration. 2014;87(1):18-25. doi: 10.1159/000346646. Epub 2013 Apr 10. PMID 23594795